CLINICAL TRIAL: NCT03997344
Title: Veterans Nature Therapy: A Pilot Randomized Trial of Hiking for Veterans With PTSD
Brief Title: Veterans Nature Therapy (Vet Hike)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Recreational Equipment, Inc. (REI) (Unknown)
Responsible Party: Principal Investigator, Gregory Bratman, Assistant Professor: College of the Environment, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006745
Record Dates: First submitted 2019-06-12; First posted 2019-06-25 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Posttraumatic Stress Disorders
Keywords: posttraumatic stress disorders; randomized controlled trial; pilot study; feasibility; nature; physical activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature hiking (Experimental): Group hikes in a natural setting (e.g., park, wilderness area)
  Interventions: Behavioral: Group nature hikes
- Urban hikes (Active Comparator): Group hikes in a urban setting (e.g., downtown area)
  Interventions: Behavioral: Group urban hikes

INTERVENTIONS:
Behavioral: Group nature hikes — Six group nature hikes will be offered once every other week. Total duration of intervention is 12 weeks. Hikes will be co-lead by two experienced hike leaders.
  Other Names: Nature hikes
  Arms: Nature hiking
Behavioral: Group urban hikes — Six group urban hikes will be offered once every other week. Total duration of intervention is 12 weeks. Hikes will be co-lead by two experienced hike leaders.
  Other Names: Urban hikes
  Arms: Urban hikes

SUMMARY:
This pilot study evaluates the feasibility of conducting a study to evaluate the impact of nature exposure/hiking in groups on symptoms of posttraumatic stress disorder in Veterans. Participants will be randomized to one of two groups: 1) nature hikes and 2) urban hikes.

DETAILED DESCRIPTION:
Objectives and hypothesis: Posttraumatic stress disorder (PTSD) is a tragically common problem among US Military Veterans. Current treatment options for PTSD are not uniformly effective and dropout rates are high. Treatment approaches that are evidence-based, effective, and acceptable to Veterans are needed. Nature therapy is a promising, low-cost intervention, yet there are few rigorous studies that have evaluated it as a therapeutic intervention in Veterans with PTSD.

The specific aims of this study are to lay the ground work for a full-scale study by assessing the feasibility and acceptability of: i) recruitment, screening, and data collection methods; and ii) the nature hiking and urban hiking control group interventions. The investigators hypothesize that the interventions will be feasible and the recruitment, screening, and data collection methods will be acceptable.

Key eligibility criteria for this two-arm pilot randomized controlled trial include being a Veterans with PTSD, physical fitness/ability sufficient to walk for at least 2 hours, and willingness to complete assessments. Eligible individuals will be randomized to one of two groups: 1) nature hiking group, 2) urban hiking group. The investigators will enroll up to 60 individuals, to randomize up to 15 participants per group. Note that the number enrolled and randomized are not expected to be the same since he investigators anticipate some individuals who enroll will be determined not to be eligible based on responses to the baseline questionnaire. Individuals randomized to groups 1 or 2 will be invited to participate in six hikes of 2-4 hours in duration, over approximately 12 weeks. Individuals will be asked to complete questionnaires at baseline and weekly for 12 weeks, and then again at 24 weeks. The primary outcomes for this study relate to feasibility and acceptability. The investigators will collect information on time to recruit the sample, retention and survey completion at each time point, and attendance at hikes. A secondary aim is to ascertain changes in PTSD symptoms (which will serve as the primary outcome of the full-scale trial), secondary outcomes (e.g., quality of life) and mediators of the intervention, including factors such as depression, perceived stress, affect, loneliness, anxiety, social connectedness, rumination, and nature connection.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Military Veteran;
* Active PTSD symptoms based on the PCL-5;
* No diagnosis of schizophrenia, bipolar disorder, or other psychotic disorders (based on self-report);
* Low risk of suicide (based on responses to the MINI Suicidal module);
* No inpatient admission in last 3 months (based on self-report);
* No current alcohol disorder/dependence (based on having a score<16 on the 10-item self-administered AUDIT questionnaire);
* No evidence of drug-related problems (based on having a score <3 on the DAST-10)
* Capable of safely participating in hikes as evidenced by no "yes's" on the Physical Activity Readiness Questionnaire (or approval of their primary care physician) and individual assertion that they can walk at least 2 hours at an easy to moderate effort with breaks;
* Willing to be randomized to one of two groups and complete all study procedures;
* Able to provide written informed consent to participate.

Exclusion Criteria:

* Schizophrenia, bipolar disorder or other psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Time to recruit the sample
Recruitment | Baseline
  Percentage of individuals contacted who are randomized
Retention | 12-week follow-up
  Percentage of participants that complete assessments

SECONDARY OUTCOMES:
PTSD symptoms | Baseline and 6-, 12-, 24-week follow-ups
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), 20 items, range 0-80; summed; higher = greater PTSD
Quality of life/well-being: Satisfaction with Life Scale | Baseline and 6-, 12-, 24-week follow-ups
  Satisfaction with Life Scale; 5-items, range 5-35; summed; higher = greater life satisfaction
Depression | Baseline and 6-, 12-, 24-week follow-ups
  Personal Health Questionnaire Depression Scale (PHQ-8); 8-items, range 3-24; summed; higher = greater depression
Perceived stress | Baseline and 6-, 12-, 24-week follow-ups
  Perceived Stress Scale 4 (PSS-4); 4-items, range 0-16; summed; higher = greater stress
Social connectedness | Baseline and 6-, 12-, 24-week follow-ups
  4-item Social Connectedness Scale; 4-items, range 4-28; summed; higher = greater connection to group
Rumination | Baseline and 6-, 12-, 24-week follow-ups
  State rumination- Rumination Reflection Questionnaire 12-items, range 5-60; summed; higher = greater rumination

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Littman, PhD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Derived] Littman AJ, Bratman GN, Lehavot K, Engel CC, Fortney JC, Peterson A, Jones A, Klassen C, Brandon J, Frumkin H. Nature versus urban hiking for Veterans with post-traumatic stress disorder: a pilot randomised trial conducted in the Pacific Northwest USA. BMJ Open. 2021 Sep 23;11(9):e051885. doi: 10.1136/bmjopen-2021-051885. PMID 34556516